CLINICAL TRIAL: NCT07160478
Title: Effectiveness of the Soc la Lola School Health Education Program on Beliefs and Knowledge About Musculoskeletal Pain Management in 8-11-Year-Old Primary School Students: Randomized Controlled Trial
Brief Title: Effectiveness of Health Education Program on Musculoskeletal Pain Management in Primary School Students
Acronym: LOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Clara Bergé Ortínez, Principal Investigator, Associate Professor at the University of Lleida, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SocLaLola_ULleida
Record Dates: First submitted 2025-08-17; First posted 2025-09-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Child, Only; Musculoskeletal Pain; Chronic Pain; School Health; Sedentary Behaviors; Health Education
Keywords: pain beliefs; pain education; children; muskuloskeletal pain; Fear-Avoidance; sedentary behaviors; Musculoskeletal pain prevention; primary school; School health program; pain science education
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Sedentary Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: After completing a pilot study, a clinical trial has been designed to evaluate an educational program aimed at preventing musculoskeletal pain in school-aged children. A total of 82 students will be divided into two groups: an intervention group (n = 42), which will participate in the new program 'SocLaLola' incorporating pain science education, and a control group (n = 40), which will follow a conventional sedentary lifestyle prevention program.
  Both sessions will be delivered by physiotherapists and will last between 45 and 60 minutes. Evaluations will be conducted immediately after the sessions and again six months later to assess the impact of the program on fear-avoidance beliefs regarding physical activity and on pain science knowledge.
Who Masked: Outcomes Assessor
Masking Description: Due to the educational nature of the intervention, it was not possible to blind participants or the physiotherapists delivering the sessions, as they were aware of the content assigned to their group. However, several procedures were implemented to ensure single-blind conditions and minimize potential bias:
  * The same physiotherapist delivered the educational sessions for both the intervention and control groups, ensuring consistency in delivery style.
  * A different member of the research team was responsible for distributing and collecting the evaluation questionnaires, reducing direct interaction between the educator and the assessment process.
  * Data analysis was conducted by an evaluator blinded to group allocation.
  * Only the principal investigator had access to the encrypted list linking participant codes to personal identifiers.
  * All questionnaires and records were pseudonymized using unique alphanumeric codes to preserve confidentiality and ensure data protection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SocLaLola Program (Experimental): Combines an explanation with the comic-based story SocLaLola to teach basic concepts of pain science education and sedentary behavior prevention in an engaging and age-appropriate way.
  Interventions: Other: School Health Program
- Stop Sedentary Behavior (Active Comparator): Delivers audiovisual materials focusing exclusively on sedentary behavior prevention, without content related to pain science education.
  Interventions: Other: School Health Program

INTERVENTIONS:
Other: School Health Program — Health education interventions of approximately 60 minutes that include a conceptual presentation and a practical component.

SUMMARY:
Musculoskeletal pain during childhood can negatively affect school attendance, physical activity, and social participation. This study will evaluate the effectiveness of the school-based health education program 'SocLaLola', which uses a comic-based narrative to introduce children to pain science concepts and promote healthy lifestyle habits. The intervention will be compared with a standard program focused on sedentary behavior prevention. Students aged 8 to 11 years from two primary schools will participate. The primary objective is to determine whether SocLaLola is more effective than the comparison program in improving children's knowledge about pain and in reducing fear-avoidance beliefs related to physical activity.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the effectiveness of the 'SocLaLola' school-based health education program compared with a sedentary lifestyle prevention program in modifying pain-related beliefs and knowledge among children aged 8 to 11 years. The primary outcomes are improvements in pain science knowledge and reductions in fear-avoidance beliefs toward physical activity.

Participants will be recruited from schools participating in the Catalan Board of Physiotherapists' School Health Program. Two primary schools will take part, each contributing two fourth-grade classes. Randomization will be performed at the class level, with classes within each school allocated to either the intervention group (SocLaLola Program) or the control group (Stop Sedentarism Program) using an online random assignment tool. This procedure ensured blocked randomization by school.

Both interventions will be delivered by trained physiotherapists in a single 45-60 minute session. The SocLaLola program combines pain science education with strategies to reduce sedentary behavior, presented through a comic-based narrative. The control group will receive audiovisual materials focusing exclusively on sedentary behavior.

Assessments will be conducted at baseline, immediately after the session, and at six months. Data collection and analysis will follow a single-blind design. Ethical approval for the study was obtained from the Research Ethics Committee of the Catalan Board of Physiotherapists (CER CFC).

ELIGIBILITY:
Inclusion criteria:

* Boys and girls from 8 to 11 years old.
* Attend the 3rd or 4th grade of primary education.
* Students from selected schools participating in the CFC project.
* Their parents or legal guardians have signed the informed consent

Exclusion criteria:

* Does not meet one or more inclusion criteria.
* Does not demonstrate reading comprehension in Catalan or Spanish.
* Does not wish to participate.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Neuroscience Knowledge (COPAQ) Score | At baseline (before intervention), immediately after intervention (same day), and at 6 months follow-up
  Change in pain neuroscience knowledge will be assessed using the validated Catalan version of the COnocimientos sobre el PAin Questionnaire (COPAQ) for children. The instrument contains 15 items with response options: true, false, or don't know. Total scores range from 0 to 15, with higher scores indicating greater knowledge of pain science.

SECONDARY OUTCOMES:
Change in Fear-Avoidance Beliefs Regarding Physical Activity (FABQ-PA) Score | At baseline (before intervention), immediately after intervention (same day), and at 6 months follow-up)
  Change in fear-avoidance beliefs will be assessed using the short Spanish version of the Fear-Avoidance Beliefs Questionnaire - Physical Activity subscale (FABQ-PA), adapted for children. The scale includes 5 items rated on a Likert scale from 0 (completely disagree) to 6 (completely agree). Total scores range from 0 to 24, with higher scores indicating greater fear-avoidance beliefs. A score above 14 is considered high fear-avoidance.
Association Between Sociodemographic Factors and Changes in Outcome Scores | At baseline (before intervention), immediately after intervention (same day), and at 6 months follow-up
  Sociodemographic variables (age, gender, school, and reported musculoskeletal pain in household members during the past three months) will be collected and analyzed as potential modifiers of changes in FABQ-PA and COPAQ scores over time.
Children's Perceived Learning After the Educational Session | Immediately after intervention (same day)
  Students will respond to the open-ended question "What do you think you learned from today's physiotherapist session?" immediately following the intervention. Qualitative responses will be analyzed thematically to explore perceived knowledge acquisition and engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bergé, MSc, PT, Principal Investigator — Universitat de Lleida
Locations (1):
- University of Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in this trial will be shared in de-identified form. Specifically, the datasets will include socio-demographic variables (age, sex, school, cohabitant pain history), responses to the Fear-Avoidance Beliefs Questionnaire (FABQ-PA), responses to the Conceptualization of Pain Questionnaire (COPAQ), and answers to the open-ended post-intervention question. All data will be pseudonymized with unique alphanumeric codes, ensuring that no personally identifiable information will be disclosed. Study protocol, statistical analysis plan, and informed consent templates will also be made available to support secondary analyses. Access to the data will require a justified request and approval by the principal investigator, and data will be shared through secure institutional repositories in accordance with ethical guidelines and data protection regulations (GDPR).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD and supporting documents (Study Protocol, SAP, ICF) will be available beginning 12 months after publication of the primary results and will remain accessible for a period of 5 years through secure institutional repositories, upon reasonable request and approval by the principal investigator.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (Study Protocol, Statistical Analysis Plan, and Informed Consent Form) will be accessible to qualified researchers affiliated with academic institutions or health research organizations, for the purpose of scientific research related to pain science education, musculoskeletal health, or school-based interventions. Access will be granted upon submission of a justified research proposal, review and approval by the principal investigator, and signature of a data access agreement. Data will be shared through secure institutional repositories in accordance with ethical standards and data protection regulations (GDPR).
URL: https://repositori.udl.cat/

REFERENCES:
- [Background] Kisling S, Claus BB, Stahlschmidt L, Wager J. The efficacy of an educational movie to improve pain and dysfunctional behavior in school children: A randomized controlled trial. Eur J Pain. 2021 Aug;25(7):1612-1621. doi: 10.1002/ejp.1777. Epub 2021 May 5. PMID 33949051
- [Background] Louw A, Landrus R, Podolak J, Benz P, DeLorenzo J, Davis C, Rogers A, Cooper K, Louw C, Zimney K, Puentedura EJ, Landers MR. Behavior Change Following Pain Neuroscience Education in Middle Schools: A Public Health Trial. Int J Environ Res Public Health. 2020 Jun 23;17(12):4505. doi: 10.3390/ijerph17124505. PMID 32585914
- [Background] Kedra A, Plandowska M, Kedra P, Czaprowski D. Physical activity and low back pain in children and adolescents: a systematic review. Eur Spine J. 2021 Apr;30(4):946-956. doi: 10.1007/s00586-020-06575-5. Epub 2020 Aug 26. PMID 32845380
- [Background] Huguet A, Tougas ME, Hayden J, McGrath PJ, Stinson JN, Chambers CT. Systematic review with meta-analysis of childhood and adolescent risk and prognostic factors for musculoskeletal pain. Pain. 2016 Dec;157(12):2640-2656. doi: 10.1097/j.pain.0000000000000685. PMID 27525834